CLINICAL TRIAL: NCT00003065
Title: Phase II Investigation of Topotecan and Taxol in Patients With Recurrent/Metastatic Cancer of the Cervix
Brief Title: Topotecan and Paclitaxel in Treating Patients With Recurrent or Metastatic Cancer of the Cervix
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Herbert Irving Comprehensive Cancer Center (Other)
Organization: National Cancer Institute (NCI) (NIH)
Purpose: Treatment
Other Study IDs: CDR0000065736; CPMC-IRB-7919; NCI-V97-1324
Record Dates: First submitted 1999-11-01; First posted 2003-01-27 (Estimated); Last update posted 2014-01-06 (Estimated); Status verified 2003-09

CONDITIONS: Cervical Cancer
Keywords: recurrent cervical cancer; stage IVB cervical cancer; stage IVA cervical cancer; cervical squamous cell carcinoma; cervical adenocarcinoma
MeSH Terms: conditions — Uterine Cervical Neoplasms | interventions — Filgrastim; Paclitaxel; Topotecan

INTERVENTIONS:
Biological: filgrastim
Drug: paclitaxel
Drug: topotecan hydrochloride

SUMMARY:
RATIONALE: Drugs used in chemotherapy use different ways to stop tumor cells from dividing so they stop growing or die. Combining more than one drug may kill more tumor cells.

PURPOSE: Phase II trial to study the effectiveness of topotecan and paclitaxel in treating patients who have recurrent or metastatic cancer of the cervix.

DETAILED DESCRIPTION:
OBJECTIVES:

* Determine the response, time to progression, disease free survival, and overall survival of patients with recurrent and/or metastatic cancer of the cervix treated with a combination of topotecan and paclitaxel.
* Determine the feasibility and toxicity of this regimen in these patients.

OUTLINE: Patients receive paclitaxel IV over 3 hours on day 1 and topotecan IV over 30 minutes on days 1-5. Filgrastim (G-CSF) is administered on days 6-14. Treatment repeats every 21 days for a minimum of 2 courses in the absence of disease progression or unacceptable toxicity.

Patients are followed every 3 weeks.

PROJECTED ACCRUAL: A total of 25 patients will be accrued for this study within 2 years.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Histologically confirmed recurrent, persistent or metastatic cervical carcinoma (squamous or adenocarcinoma), with no potentially curative standard treatment
* Measurable disease or evaluable disease

PATIENT CHARACTERISTICS:

Age:

* 18 to physiological 60

Performance status:

* ECOG 0-2

Life expectancy:

* Greater than 2 months

Hematopoietic:

* WBC greater than 3000/mm3
* Platelet count greater than 100,000/mm3

Hepatic:

* Bilirubin less than 1.5 times normal
* SGOT/SGPT less than 1.5 times normal

Renal:

* BUN less than 1.5 times normal
* Creatinine less than 1.5 times normal
* Creatinine clearance greater than 50 mL/min

Other:

* Ineligible for other high priority national or institutional study
* Not pregnant or nursing
* HIV negative
* No prior malignancy except nonmelanoma skin cancer
* No serious medical or psychiatric illness preventing treatment or informed consent

PRIOR CONCURRENT THERAPY:

Biologic therapy:

* Not specified

Chemotherapy:

* Greater than 4 weeks since prior chemotherapy
* No greater than 2 prior chemotherapy regimens
* No prior taxane or camptothecin

Endocrine therapy:

* No concurrent hormonal therapy except that required for nondisease related conditions (e.g., insulin for diabetes)

Radiotherapy:

* Greater than 4 weeks since prior radiation therapy
* No concurrent radiation therapy

Surgery:

* Greater than 4 weeks since prior surgery

Ages: 18 Years to 60 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 25 (Estimated)
Dates: Start 1997-01; Study Completion 2004-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Amy D. Tiersten, MD, Study Chair — Herbert Irving Comprehensive Cancer Center
Locations (1):
- Herbert Irving Comprehensive Cancer Center at Columbia University, New York, New York, United States

REFERENCES:
- [Result] Tiersten AD, Selleck MJ, Hershman DL, Smith D, Resnik EE, Troxel AB, Brafman LB, Shriberg L. Phase II study of topotecan and paclitaxel for recurrent, persistent, or metastatic cervical carcinoma. Gynecol Oncol. 2004 Feb;92(2):635-8. doi: 10.1016/j.ygyno.2003.11.019. PMID 14766258